CLINICAL TRIAL: NCT04182165
Title: Non-Contact Monitoring of Subjects With an Optical Device: A Pilot Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ContinUse Biometrics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CUBX-08
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-01

CONDITIONS: Usability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects measured by the study staff (Experimental): Subjects measured by the study staff via the investigational device at the hospital (up to 50 subjects).
  Interventions: Device: Gili BioSensor System/ Gili Pro X BioSensor System
- Subjects measuring themselves autonomously (Experimental): Subjects measuring themselves autonomously with the investigational device at their homes (up to 10 subjects from the first arm).
  Interventions: Device: Gili BioSensor System/ Gili Pro X BioSensor System

INTERVENTIONS:
Device: Gili BioSensor System/ Gili Pro X BioSensor System — Usability study

SUMMARY:
This is a single-center, prospective study in subjects visiting TASMC for various indications.

This study will be divided into two arms:

First Arm - Subjects measured by the study staff via the investigational device at the hospital (up to 50 subjects).

Second Arm - subjects measuring themselves autonomously with the investigational device at their homes (up to 10 subjects from the first arm).

Hence, total number of subjects for the study will be up to N=50. All subjects will be enrolled to the study only after signing an informed consent form.

Specifically for the second arm, subjects will undergo proper training by the sponsor's representatives prior to being discharged from the hospital. Training will focus on proper operation of the device, which is also designed for autonomous use in a simple and user-friendly manner. Subjects will be asked to monitor themselves periodically for a duration of up to a week. Ongoing support will be provided by the sponsor upon subject request, either by phone, or on-premise via a dedicated support team.

For both arms, device users (either study staff in first arm or subjects in the second arm) will be requested to answer questionnaires in order to assess usability with the investigational device. In both cases, a dedicated sponsor representative will observe the users to gather objective usability data, and aid in the questionnaire filling process.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age, male or female
* Hemodynamically stable as assessed by the investigator

Exclusion Criteria:

* Inability to comply with study protocol as assessed by the study staff (e.g. currently suffering from tremors, afraid of using tech-based devices etc.)
* Inability to provide informed consent
* Parallel participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Questionnaires assessed by SUS score and answered by the study staff. | During the procedure
Questionnaires assessed by SUS score and answered by the enrolled study subjects. | During the procedure
Measurement of vital signs (Heart rate/ Respiratory rate) acquired via the investigational device along with de-identified subject medical data. | During the procedure

SECONDARY OUTCOMES:
Safety assessed by AE/SAE | During the procedure
  The Gili System functions without physical contact with the inspected subject and is designed as a class 1 laser product (fully eye safe). Consequently, we do not expect any safety issues. At the same time, any AEs occurring during both trial stages will be recorded in the CRF.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center (TASMC), Tel Aviv, Israel